CLINICAL TRIAL: NCT00390208
Title: A Prospective Masked Pilot Study Comparing Group 1 Triple Therapy - PDT Plus IVD and Intravitreal Ranibizumab Versus Group 2 Monotherapy - Intravitreal Ranibizumab Alone.
Brief Title: Triple Therapy - PDT Plus IVD and Intravitreal Ranibizumab Versus Lucentis Monotherapy to Treat Age-Related Macular Degeneration
Acronym: PDEX
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bay Area Retina Associates (Other)
Collaborators: QLT Inc. (Industry)
Responsible Party: Subhransu K. Ray, M.D., Ph.D., Bay Area Retina Associates
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PDEX
Record Dates: First submitted 2006-10-17; First posted 2006-10-19 (Estimated); Last update posted 2010-05-27 (Estimated); Status verified 2010-05

CONDITIONS: Age Related Macular Degeneration
Keywords: Macular Degeneration; Degenerative changes in the macula lutea of the retina.; Maculopathy, Age-Related; Age-Related Maculopathies; Age-Related Maculopathy; Maculopathies, Age-Related; RETINAL DEGENERATION; ARMD; AMD; Lucentis; Visudyne; Photodynamic Therapy; Verteporfin; Ranibizumab; Intravitreal Dexamethasone
MeSH Terms: conditions — Macular Degeneration; Retinal Degeneration | interventions — Ranibizumab; Dexamethasone; Verteporfin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1 (Other): Combination triple therapy of Lucentis, Dexamethasone and Visudyne Therapy
  Interventions: Drug: ranibizumab, dexamethasone and verteporfin
- Group 2 (Other): Monotherapy: One 0.5 mg intravitreal Ranibizumab injection
  Interventions: Drug: Ranibizumab

INTERVENTIONS:
Drug: ranibizumab, dexamethasone and verteporfin — One 500 microgram dose (0.05cc) intravitreal dexamethasone (10 mg/ml vial) in combination with Visudyne Photodynamic Therapy and 0.5 mg intravitreal Ranibizumab injection on the same day.
  Arms: Group 1
Drug: Ranibizumab — One 0.5 mg intravitreal Ranibizumab injection
  Arms: Group 2

SUMMARY:
The purpose of this study is to compare triple therapy using Photodynamic therapy, intravitreal Dexamethasone and intravitreal Ranibizumab injections versus monotherapy with intravitreal Ranibizumab alone for the treatment of Age-Related Macular Degeneration.

DETAILED DESCRIPTION:
This is a twelve month Phase II prospective masked study comparing Group 1 triple therapy: Same day combination therapy with PDT, 500 microgram dose (0.05cc) intravitreal dexamethasone injection (10mg/ml vial), and a single 0.5 mg intravitreal Ranibizumab injection. This will be compared to Group 2 monotherapy: one intravitreal injection of 0.5 mg Lucentis given every four weeks on a set dosing schedule. Sixty consecutive patients will be enrolled into this clinical trial utilizing the current standard of care guidelines as used at Bay Area Retina Associates. Angiography, fundus photography will be performed at the initial visit and quarterly follow-up visits. Only OCT testing will be performed at all other follow-up visits. Both groups will be re-evaluated for safety at 12 and 24 months.

Group 1 Following the initial treatment, all future re-treatments with Lucentis will be determined on a PRN basis. The decision will be based on clinical examination and imaging evidence of lesion activity. Any evidence of subretinal fluid or cystoid edema on OCT or clinical examination, or evidence of leakage on angiogram will result in re-treatment. If after three consecutive Ranibizumab injections in Group 1, there is any evidence of lesion recurrence or growth of the neovascular membrane associated with visual decline or persistent subretinal fluid, the patient will be treated with repeat PDT/IVD/Lucentis The decision to retreat Group 1 with ranibizumab at each monthly follow-up visit will be dependent on clinical exam, OCT measurements or angiographic findings as documented below.

Group 2 Subjects will receive one intravitreal injection of 0.5 mg Lucentis every four weeks until week 48 or as indicated on the FDA approval label.

ELIGIBILITY:
Inclusion Criteria:

* Best Corrected Visual Acuity using ETDRS Charts between 20/32 and 20/400 (Snellen Equivalent) in the study eye with evidence of neovascular ARMD.

(Only one eye will be eligible for study. If both eyes are eligible, the one with the better visual acuity will be selected for treatment unless, based on medical reasons, the investigator deems the other eye to be more appropriate for treatment and study.)

* All lesion subtypes will be enrolled with the following criteria

  * Predominantly classic:
* Classic lesion greater than 50% of the total lesion area
* Lesion must be less than 12 disc areas

  * Minimally classic or occult:
* CNVM must be greater than or equal to 50% of the total lesion size.
* There must be some evidence of recent disease progression (heme, vision loss, recent lesion growth on FA)
* Lesion size must be less than 12 disc areas.

  * Occult:
* Lesions must show recent activity progression with respect to vision, subretinal hemorrhage or subretinal fluid
* Less than 12 disc areas in total size
* Signed informed consent
* Age greater than or equal to 50 years

Exclusion Criteria:

* Pigment epithelial detachment greater than 50% of the total lesion size
* Previous treatment for ARMD in the study eye
* Previous intravitreal drug delivery in the study eye
* History of vitrectomy in the study eye
* Fibrosis or atrophy involving the center of the fovea in the study eye
* Neovascular membrane from any other concurrent retinal disease such as high myopia (SER > -8D), histoplasmosis or other ocular inflammatory disease.
* Known history of glaucoma and on more than one topical medication
* History of glaucoma filtering surgery in the study eye
* History of corneal transplant in the study eye
* Patients with co-existing macular disease such as diabetic macular edema
* Active intraocular inflammation in the study eye
* History of allergy to fluorescein not amenable to treatment
* Inability to comply with study or follow up procedures

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2006-08; Primary Completion 2008-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Visual Acuity: Change in visual acuity by 15 or more ETDRS letters at 6 and 12 months. Non-inferiority as compared to the triple therapy arm will serve to determine efficacy for the purposes of this pilot trial. | one year

SECONDARY OUTCOMES:
Lesion size | one year
Lesion leakage | one year
OCT measurement of macular thickness, subretinal fluid and cystoid edema | one year
Total number of treatments required | one year
Timing of visual improvement after initiation of therapy | one year

CONTACTS AND LOCATIONS:
Overall Officials: Subhransu K Ray, M.D., Ph.D., Principal Investigator — Bay Area Retina Associates
Locations (4):
- United States (4):
  - Bay Area Retina Associates, Castro Valley, California
  - Bay Area Retina Associates, Walnut Creek, California
  - Georgia Retina, Riverdale, Georgia
  - Retina Vitreous Associates, Toledo, Ohio

REFERENCES:
- [Background] Bressler NM, Arnold J, Benchaboune M, Blumenkranz MS, Fish GE, Gragoudas ES, Lewis H, Schmidt-Erfurth U, Slakter JS, Bressler SB, Manos K, Hao Y, Hayes L, Koester J, Reaves A, Strong HA; Treatment of Age-Related Macular Degeneration with Photodynamic Therapy (TAP) Study Group. Verteporfin therapy of subfoveal choroidal neovascularization in patients with age-related macular degeneration: additional information regarding baseline lesion composition's impact on vision outcomes-TAP report No. 3. Arch Ophthalmol. 2002 Nov;120(11):1443-54. doi: 10.1001/archopht.120.11.1443. PMID 12427056
- [Background] VEGF Inhibition Study in Ocular Neovascularization (V.I.S.I.O.N.) Clinical Trial Group; D'Amico DJ, Masonson HN, Patel M, Adamis AP, Cunningham ET Jr, Guyer DR, Katz B. Pegaptanib sodium for neovascular age-related macular degeneration: two-year safety results of the two prospective, multicenter, controlled clinical trials. Ophthalmology. 2006 Jun;113(6):992-1001.e6. doi: 10.1016/j.ophtha.2006.02.027. Epub 2006 Apr 27. PMID 16647134
- [Background] Avery RL, Pieramici DJ, Rabena MD, Castellarin AA, Nasir MA, Giust MJ. Intravitreal bevacizumab (Avastin) for neovascular age-related macular degeneration. Ophthalmology. 2006 Mar;113(3):363-372.e5. doi: 10.1016/j.ophtha.2005.11.019. Epub 2006 Feb 3. PMID 16458968
- [Background] Edelman JL, Lutz D, Castro MR. Corticosteroids inhibit VEGF-induced vascular leakage in a rabbit model of blood-retinal and blood-aqueous barrier breakdown. Exp Eye Res. 2005 Feb;80(2):249-58. doi: 10.1016/j.exer.2004.09.013. PMID 15670803
- [Background] Spaide RF, Sorenson J, Maranan L. Photodynamic therapy with verteporfin combined with intravitreal injection of triamcinolone acetonide for choroidal neovascularization. Ophthalmology. 2005 Feb;112(2):301-4. doi: 10.1016/j.ophtha.2004.08.012. PMID 15691567
- [Background] Shah GK, Stein JD, Sharma S, Sivalingam A, Benson WE, Regillo CD, Brown GC, Tasman W. Visual outcomes following the use of intravitreal steroids in the treatment of postoperative endophthalmitis. Ophthalmology. 2000 Mar;107(3):486-9. doi: 10.1016/s0161-6420(99)00139-6. PMID 10711885
- [Background] Tamura H, Miyamoto K, Kiryu J, Miyahara S, Katsuta H, Hirose F, Musashi K, Yoshimura N. Intravitreal injection of corticosteroid attenuates leukostasis and vascular leakage in experimental diabetic retina. Invest Ophthalmol Vis Sci. 2005 Apr;46(4):1440-4. doi: 10.1167/iovs.04-0905. PMID 15790913
- [Background] Chalam KV, Malkani S, Shah VA. Intravitreal dexamethasone effectively reduces postoperative inflammation after vitreoretinal surgery. Ophthalmic Surg Lasers Imaging. 2003 May-Jun;34(3):188-92. PMID 12757090
- [Background] Blankenship GW. Evaluation of a single intravitreal injection of dexamethasone phosphate in vitrectomy surgery for diabetic retinopathy complications. Graefes Arch Clin Exp Ophthalmol. 1991;229(1):62-5. doi: 10.1007/BF00172263. PMID 2004725
- [Background] Schmidt-Erfurth U, Schlotzer-Schrehard U, Cursiefen C, Michels S, Beckendorf A, Naumann GO. Influence of photodynamic therapy on expression of vascular endothelial growth factor (VEGF), VEGF receptor 3, and pigment epithelium-derived factor. Invest Ophthalmol Vis Sci. 2003 Oct;44(10):4473-80. doi: 10.1167/iovs.02-1115. PMID 14507895
- [Background] Wenzel A, Grimm C, Seeliger MW, Jaissle G, Hafezi F, Kretschmer R, Zrenner E, Reme CE. Prevention of photoreceptor apoptosis by activation of the glucocorticoid receptor. Invest Ophthalmol Vis Sci. 2001 Jun;42(7):1653-9. PMID 11381074
- [Background] Augustin AJ, Schmidt-Erfurth U. Verteporfin and intravitreal triamcinolone acetonide combination therapy for occult choroidal neovascularization in age-related macular degeneration. Am J Ophthalmol. 2006 Apr;141(4):638-45. doi: 10.1016/j.ajo.2005.11.058. PMID 16564797
- [Background] Nicolo M, Ghiglione D, Lai S, Nasciuti F, Cicinelli S, Calabria G. Occult with no classic choroidal neovascularization secondary to age-related macular degeneration treated by intravitreal triamcinolone and photodynamic therapy with verteporfin. Retina. 2006 Jan;26(1):58-64. doi: 10.1097/00006982-200601000-00010. PMID 16395140
- [Background] Spaide RF, Laud K, Fine HF, Klancnik JM Jr, Meyerle CB, Yannuzzi LA, Sorenson J, Slakter J, Fisher YL, Cooney MJ. Intravitreal bevacizumab treatment of choroidal neovascularization secondary to age-related macular degeneration. Retina. 2006 Apr;26(4):383-90. doi: 10.1097/01.iae.0000238561.99283.0e. PMID 16603955
- [Background] Maturi RK, Bleau LA, Wilson DL. Electrophysiologic findings after intravitreal bevacizumab (Avastin) treatment. Retina. 2006 Mar;26(3):270-4. doi: 10.1097/00006982-200603000-00003. PMID 16508425
- [Background] Manzano RP, Peyman GA, Khan P, Kivilcim M. Testing intravitreal toxicity of bevacizumab (Avastin). Retina. 2006 Mar;26(3):257-61. doi: 10.1097/00006982-200603000-00001. PMID 16508423
- See also: Study Sponsor website — http://www.bayarearetina.com